CLINICAL TRIAL: NCT06877819
Title: Additional Effects of Motor Imagery Technique Along With Task Oriented Trunk Control Training on Postural Control And Mobility In Stroke Patients
Brief Title: Additional Effects of Motor Imaginary Technique Along With Task Oriented Trunk Control Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/MS-PT/02027 Minahil Butt
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Stroke
Keywords: balance; mobility; motor imaginary; posture; trunk
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Imaginary alongwith Task Oriented Training (Experimental): patient will first imagine task task-based based activities with closed eyes while listening to the audio using headphones, this will be followed by practical implication of same tasks and coventional physiotherapy.
  Interventions: Other: Motor Imaginary Technique alongwith task-oriented training
- Task Oriented Training (Active Comparator): patient will be asked to perform task based activities followed by conventional physiotherapy
  Interventions: Other: Task Oriented Training

INTERVENTIONS:
Other: Motor Imaginary Technique alongwith task-oriented training — Motor imaginary technique followed by task oriented trunk control training alongwith conventional physiotherapy.Frequency: 10- 15 reps 4 times/week for 8 consecutive weeks. Time for each session will be 60 mins. First of all task based exercises will be assumed by patient. To make imaginations more strong an audio demonstration of each exercise will be recorded by therapist and will be administered to patients hearing via headphones. This will make it easy for patients to assume as they are performing theses exercises in their head. Motor imagination will be followed by practical performance of same tasks. The experimental group will receive motor imagery technique for 15 minutes followed by task-specific training for 45minutes along with conventional physiotherapy to improve postural control and balance in stroke patients. .
  Arms: Motor Imaginary alongwith Task Oriented Training
Other: Task Oriented Training — Control group will receive task oriented trunk control training exercises followed by conventional physiotherapy. .Frequency: 10- 15 reps 4 times/week for 8 consecutive weeks. Time for each session will be 60 mins.
  Arms: Task Oriented Training

SUMMARY:
The aim of this randomized controlled trial is determine additional effects of motor imagery technique along with task oriented training on trunk control, posture, balance and mobility.

DETAILED DESCRIPTION:
Stroke has been classified as leading cause of death and disability. Mild to severe disruption on physical and cognitive functions may occur in stroke patients. Lack of motor control, muscle control, sensations, balance commonly develop after stroke. Motor dysfunctions result in body paralysis, paresis, stiffness, decrease range of motion, thereby limiting mobility, body movements hence increasing dependance in performing activities of daily living. Majority of patients of stroke face trunk and pelvis instability and asymmetry resulting in swaying posture, decreased stability, difficulty in weight shifting on affected side therefore resulting in impaired balance. One of advanced technique used in stroke patients is an active cognitive approach known as motor imagery technique (MIT). It involves mental rehearsal of simple and complex movements as per required internally in working memory of a person followed by asking patient to try practical implementation of imagined movement or task at end of each session. Thus this technique is constant reprocessing of interpretation that arise from perception of movement created in mind of a patient enhancing neural connections. In today's world intervention has been goal oriented involving task specific training i.e., repetitive practice of functional task incorporating desired movement and action during activity there by regulating nervous system re-building neural pathways through repeated practice. Task specific training enhance performance of trunk muscles by focusing on concept of function, participation and quality of life. To gain gainful effects among stroke patients, combining cognitive developmental strategy with physical goal oriented activity can be fruitful as it nourishes the concept of neuronal recruitment along with motor control development by improving trunk control, posture and balance among stroke patients. The rationale for the use of these techniques is to identify additional effects of MIT along with task oriented training on trunk control and mobility as studies conducted on trunk control using MI in past were devoid of activity based training, where as those conducted using task-oriented training lack advancement in technology. Therefore, due to dearth of empirical data on symbiotic benefits of motor imagery technique along with task oriented training leads to foundation of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sub-acute stroke (> 3 months stroke till 6 months after stroke)
* Both male and female are included.
* Patient with stage 2 of postural control on Chedoke McMaster Stroke Assessment Score.
* Patient who are able to sit without holding on to objects/people
* Patient who are able to stand for 30seconds
* Patient able to flex non-paretic shoulder upto 90 degree, without holding on to any object
* Patients with no cognitive deficits ( score > 25 on Montreal Cognitive Assessment Tool)
* Patients with moderate spasticity of upper/lower extremity (Modified Ashworth Scale Grade = 1, +1)

Exclusion Criteria

* Patients with visuo-spatial neglect.
* Patients with hearing impairment
* Hip pathologieOlder adults 60 years & aboves or any condition other than stroke interfering with trunk movements will be excluded

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Postural Assesment Scale for Stroke | 8 weeks
  it was developed in 1999 as an adaptation to fugyl-meyer scale. PASS scale is designed for stroke patient to assess and monitor postural control after stroke. Multiple studies support the predictive validity of the PASS. PASS demonstrated excellent predictive validity at 14, 30, 90 and 180 days post stroke (α=0.86-0.90), as measured using Spearman's p correlation coefficient.
  The PASS scale is composed of 2 sections of posture I.e: maintaining posture and changing a posture. it is a 4-point scale and consist a total of 12 items with total score of 36.
Trunk Impairment Scale | 8 weeks
  TIS was developed by Verheydenet. al to evaluate trunk control in stroke patients. TIS assesses static and dynamic sitting balance and trunk coordination in a sitting position. The total score for TIS ranges between 0 for a minimal performance to 23 for a perfect performance. Test/retest and interobserver reliability for the TIS total score (ICC) - 0.96 and 0.99, respectively. The 95% limits of agreement for the test/retest and interexaminer measurement error - 2/2.90, 3.68 and 2/1.84, 1.84, respectively. Cronbach alpha coefficients for internal consistency range from 0.65 to 0.89.
Berg Balance Scale | 8 weeks
  The Berg Balance Scale (BBS) is used to determine balance Impairment in elderly. population and in patients with strok . It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. The Berg Balance Scale has a high relative reliability with inter-rater reliability estimated at 0.97 (95% CI 0.96 to 0.98) and intra-rater reliability estimated at 0.98 (95% CI 0.97 to 0.99).
Functional Reach Test | 8 weeks
  In 1990 Pamela Duncan and colleagues developed Functional Reach test. It is single-task, dynamic test that is used to predict falls in older adults. This test measures the margin of stability along with the ability to measure balance during a functional task. Correlation values were 0.86 and 0.87 at two different times, with a correlation coefficient greater than 0.76 is a strong predictor of fall.
Time-Up and-Go Test | 8 weeks
  The Timed Up and Go (TUG) is a commonly used outcome measure that can assess activity limitations in the ICF model by examining the patient's ability to ambulate and perform transfers. The Timed up and Go test has excellent inter-rater correlation (ICC) = 0.99, and high intra-rater reliability (ICC = 0.99).
5 Times sit-t-To-Stand Test | 8 weeks
  5 times sit to stand test (5XSST) measures functional lower limb muscle strength and may be useful in quantifying functional change of transitional movements. The 5XSST test has excellent intra-rater reliability (intraclass correlation coefficient (ICC) range: 0.914-0.933) and excellent test-retest reliability (ICC range: 0.988-0.995) in healthy older adults.

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Nawaz Malik, PhD Rehab, Principal Investigator — Riphah International University; Minahil Butt, MS-NMPT*, Principal Investigator — Riphah International University
Locations (1):
- National Institute of Rehab Medicine, Nijaat Ambulance & Old Age Home, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No